CLINICAL TRIAL: NCT00881205
Title: A 16-week, Multicenter, Double-blind, Randomized, Placebo-controlled, Parallel Group Study to Evaluate the Efficacy of Rivastigmine Patch (10 cm²) on Cognitive Deficits in Patients With Multiple Sclerosis, Followed by a 1-year Open-label Treatment Phase
Brief Title: Rivastigmine in Multiple Sclerosis Patients With Cognitive Impairment
Acronym: EXCITING
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Termination of study due to low enrollment
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CENA713DDE18
Record Dates: First submitted 2009-04-14; First posted 2009-04-15 (Estimated); Results first posted 2012-02-24 (Estimated); Last update posted 2012-03-12 (Estimated); Status verified 2012-03

CONDITIONS: Multiple Sclerosis; Cognitive Impairment
Keywords: Multiple Sclerosis; Cognition; Rivastigmine; Patch
MeSH Terms: conditions — Multiple Sclerosis; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Rivastigmine (Experimental): Rivastigmine patch arm with the application of one 5 cm² patch, followed by an increase to the target dose of 10 cm² patch size.
  Interventions: Drug: Rivastigmine transdermal patch
- Placebo (Placebo Comparator): Placebo patch arm with the application of one 5 cm² patch, followed by an increase to the target dose of 10 cm² patch size.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rivastigmine transdermal patch — Transdermalapplication of one 5 cm² patch, followed by an increase to the target dose of 10 cm² patch size. All patches are round, beige in color.
  Arms: Rivastigmine
Drug: Placebo — Transdermal application of one 5 cm² patch, followed by an increase to the target dose of 10 cm² patch size. Matching the size, shape and color of rivastigmine patches.
  Arms: Placebo

SUMMARY:
This study evaluated the efficacy and safety of 10 cm² rivastigmine patch vs. placebo in cognitively impaired Multiple Sclerosis (MS) patients. Primary objective was the assessment of cognition by the Selective Reminding Test (SRT) -a subtest of the brief repeatable battery (BRB) - after titration of 4 weeks and maintenance of 12 weeks. This double-blind period was followed by a 52-week open-label treatment phase to assess long-term safety of rivastigmine patch in these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent to participate in the trial
2. Males and females between 18 and 55 years of age;
3. Definite diagnosis of multiple sclerosis as defined by 2005 revised McDonald criteria
4. MS-subtype: Clinical isolated syndrome (CIS), Relapsing Remitting Multiple Sclerosis (RRMS), Secondary progressive Multiple Sclerosis (SPMS);
5. Cognitive Impairment
6. Sufficient education to read, write and communicate comprehensibly

Exclusion Criteria:

1. Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer
2. Women who are pregnant or breast feeding or who are menstruating and capable of becoming pregnant and not practicing a medically approved method of contraception
3. With a physical or sensory disability that can subjectively prevent the patient from completing all study requirements
4. Patients suffering any other type of concomitant psychiatric and/or neurological disorder other than MS which is known to affect cognition (e.g. severe depressive symptoms, cerebrovascular diseases, epilepsy).
5. Patients suffering an acute relapse of MS in the previous 30 days (treated or not with intravenous or oral glucocorticoid regimens) prior to baseline.
6. With a history or current problem of drug-addiction and/or alcohol abuse.
7. Known or 'new' diagnosis of diabetes mellitus (if screening blood glucose is suspicious for diabetes [≥126 mg/dL or ≥7 mmol/L if fasting and ≥200 mg/dL or 11.1 mmol/L if random testing] a patient should be further evaluated for diabetes mellitus)
8. With a history of severe or moderate-severe cranioencephalic trauma.
9. History or presence of any intolerance or contraindication for the application of rivastigmine (or for drugs with similar chemical structures) as listed in the current Investigator's Brochure and/or SPC, i.e. severe liver insufficiency, pancreatitis, gastric ulcer, convulsions.
10. With a history in the past year or a current diagnosis of cerebrovascular disease (for instance, stroke, transient ischemic events, aneurysms).
11. Severe depressive symptoms indicated by a score of more than ≥ 14 on the MADRS at screening
12. History of malignancy of any organ system, treated or untreated, within the past 5 years whether or not there is evidence of local recurrence or metastases, with the exception of localized basal cell carcinoma of the skin

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2009-04; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (43):
- Germany (43):
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Aalen
  - Novartis Investigative Site, Abensberg
  - Novartis Investigative Site, Achim
  - Novartis Investigative Site, Alzenau in Unterfranken
  - Novartis Investigative Site, Aschaffenburg
  - Novartis Investigative Site, Bad Mergentheim
  - Novartis Investigative Site, Bayreuth
  - Novartis Investigative Site, Berlin
  - Novartis Investigative SIte, Berlin
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Böblingen
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Eisenach
  - Novartis Investigative Site, Ellwangen
  - Novartis Investigative Site, Erbach im Odenwald
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Giessen
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigational Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Itzehoe
  - Novartis Investigative Site, Kaltenkirchen
  - Novartis Investigative Site, Krefeld
  - Novartis Investigative Site, Lappersdorf
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Ludwigshafen
  - Novartis Investigative Site, Lüneburg
  - Novartis Investigative Site, Neu-Ulm
  - Novartis Investigative Site, Neuburg am Inn
  - Novartis Investigative Site, Oldenburg
  - Novartis Investigative Site, Osnabrück
  - Novartis Investigative Site, Rostock
  - Novartis Investigative Site, Stade
  - Novartis Investigative Site, Stuttgart
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Unterhaching
  - Novartis Investigative Site, Viernheim
  - Novartis Investigative Site, Wiesbaden
  - Novartis Investigative Site, Wolfratshausen

RESULTS

PARTICIPANT FLOW:
Groups:
- Rivastigmine: 5 and 10 cm² patch sizes (4,6mg/24h or 9,5mg/24h) of rivastigmine,
- Placebo: Matching the size, shape and color of rivastigmine patches.
Period: Overall Study
Arm/Group | Rivastigmine | Placebo
Started | 45 | 41
Completed | 34 | 34
Not Completed | 11 | 7
Not completed — Adverse Event | 8 | 3
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Administrative problems | 1 | 1
Not completed — Condition no longer requires drug | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rivastigmine | Placebo | Total
Number analyzed (Participants) | 43 | 38 | 81
Age Continuous [Mean (Standard Deviation); unit: years] | 44.6 (9.4) | 44.0 (7.3) | 44.3 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 20 | 43
  Male | 20 | 18 | 38

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 16 in Total Recall on the Selective Reminding Test (SRT) in the Intent to Treat (ITT) Population
Description: The Selective Reminding Test(SRT) is a test to assess verbal learning and memory. During the administration of the SRT only the examiner and the patient should be in the testing room. A list of twelve words is read aloud by the examiner at a rate of one word per two seconds. The patient is asked to recall all twelve words. Only the words that are missed on the preceding trial are given in the consecutive trial. The total score represents a sum score of 6 trials, therefore the range is from 0-72. The lower the value the worse the outcome.
Time Frame: After 16 weeks of treatment
Population: Due to low enrollment numbers study did not achieve the anticipated 80% power.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rivastigmine | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The safety population will consist of all patients that received at least one dose of study drug and had at least one post-baseline safety assessment. Patients will be analyzed according to treatment received.
Groups:
- Total Patients: Total Patients
Arm/Group | Total Patients | Rivastigmine | Placebo
Serious Adverse Events (participants affected / at risk) | 6/86 | 2/45 | 4/41
Other Adverse Events (participants affected / at risk) | 48/86 | 25/45 | 23/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Total Patients (N=86) | Rivastigmine (N=45) | Placebo (N=41)
NAUSEA (Gastrointestinal disorders) | 1 | 0 | 1
OEDEMA PERIPHERAL (General disorders) | 1 | 0 | 1
PYREXIA (General disorders) | 1 | 0 | 1
CELLULITIS (Infections and infestations) | 1 | 1 | 0
PYELONEPHRITIS (Infections and infestations) | 1 | 1 | 0
SEPSIS (Infections and infestations) | 1 | 1 | 0
DIZZINESS (Nervous system disorders) | 1 | 0 | 1
OPTIC NEURITIS (Nervous system disorders) | 1 | 0 | 1
DEPRESSION (Psychiatric disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Total Patients (N=86) | Rivastigmine (N=45) | Placebo (N=41)
VERTIGO (Ear and labyrinth disorders) | 3 | 2 | 1
DIARRHOEA (Gastrointestinal disorders) | 3 | 1 | 2
NAUSEA (Gastrointestinal disorders) | 6 | 2 | 4
VOMITING (Gastrointestinal disorders) | 3 | 2 | 1
CHILLS (General disorders) | 2 | 2 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 3 | 1 | 2
NASOPHARYNGITIS (Infections and infestations) | 7 | 6 | 1
RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 0 | 2
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
DIZZINESS (Nervous system disorders) | 2 | 0 | 2
MULTIPLE SCLEROSIS RELAPSE (Nervous system disorders) | 10 | 4 | 6
DEPRESSION (Psychiatric disorders) | 5 | 1 | 4
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2
ERYTHEMA (Skin and subcutaneous tissue disorders) | 13 | 7 | 6
PRURITUS (Skin and subcutaneous tissue disorders) | 3 | 2 | 1
RASH (Skin and subcutaneous tissue disorders) | 7 | 5 | 2
SKIN IRRITATION (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
SKIN REACTION (Skin and subcutaneous tissue disorders) | 3 | 1 | 2
HYPERTENSION (Vascular disorders) | 3 | 2 | 1

LIMITATIONS AND CAVEATS:
This study was terminated early due to low recruitment numbers. This study did not have the anticipated 80% power.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.